CLINICAL TRIAL: NCT03561402
Title: Association of Possible Biomarkers With Disease Activity in Patients Treated With Teriflunomide (Aubagio)
Brief Title: Biomarkers and Disease Activity in Patients Treated With Teriflunomide (Aubagio)
Status: Completed | Type: Observational
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, David Haegert, Professor, McGill University
Other Study IDs: GZ-2015-11483
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: biomarker; teriflunomide; activity
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Motor Activity | interventions — teriflunomide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cryopreserved peripheral blood mononuclear cells (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with active disease: From the cohort of patients receiving teriflunomide - 1 tablet (14 mg) daily, the investigators will identify patients that have active disease..
  Interventions: Drug: Teriflunomide
- Patients with stable disease: From the cohort of patients receiving teriflunomide (as above), the investigators will identify patients that have stable disease.
  Interventions: Drug: Teriflunomide

INTERVENTIONS:
Drug: Teriflunomide — Each patient will receive 1 tablet (14 mg) on a daily basis.
  Other Names: Aubagio

SUMMARY:
The study is a two-year prospective observational study of patients treated with teriflunomide. The investigators will recruit up to 75 patients at baseline, based on the estimate that approximately 20% of these patients (~ 15 patients) will have evidence of disease activity at the end of the first year of treatment with teriflunomide, as determined by clinical evaluation (relapses) and MRI activity (new T2 hyperintense lesions). The investigators will assess the expression of a putative biomarker signature consisting of toll like receptor 2(TLR2), TLR4 and chemokine receptor 1 (CCR1) on CD4 T-subsets at baseline and at intervals on treatment with teriflunomide to determine whether expression of this biomarker signature on one or more CD4 T-subsets correlates with disease activity.

DETAILED DESCRIPTION:
TITLE: Association of possible biomarkers with disease activity in patients treated with teriflunomide (Aubagio ®)

A. BACKGROUND Teriflunomide (Aubagio) is a once-daily oral immunomodulatory DMT for patients with relapsing-remitting MS (RRMS) (1). The objective of the present study is to determine whether a putative biomarker signature predicts disease activity in patients treated with teriflunomide. The investigators previously identified a 130-gene signature associated with immune activation that identified patients with MS that had rapid transition to secondary progressive MS (SPMS). From this signature, the investigators identified three genes (TLR2, TLR4 and CCR1) which had increased protein expression on naïve CD4 T-cells in these patients. The investigators also showed that mRNA for an anti-proliferation factor, termed TOB1, was downregulated in these T-cells in patients with rapid MS progression. The findings suggest, therefore, that naïve CD4 T-cell activation identifies patients with MS having a short RRMS duration (2).

For this proposal, the principal investigator suggests that various molecules involved in T-cell activation may also serve as useful biomarkers to predict treatment responses to teriflunomide.

B. STUDY OBJECTIVES

B1. Study objective and specific aims. The objective is to determine whether the T-cell activation markers that were previously identified will predict disease activity in patients treated with teriflunomide.

The specific study aims are to determine:

1. the proportion of patients pre-treatment (pre-Tx) that have altered expression of one or more candidate markers in one or more T-subsets;
2. whether expression levels of one or more of these markers in a T-subset change(s) on treatment (On-Tx) with teriflunomide;
3. whether differences in the mRNA or protein kinetics of a putative marker predicts disease activity in patients treated with teriflunomide;
4. whether expression levels of one or more target molecules, Pre-Tx or On-Tx, correlate with evidence of disease activity after one year on treatment.

C. STUDY DESIGN.

C1. Design summary. The study is a two-year prospective observational study of patients treated with teriflunomide. The investigators will recruit up to 75 patients at baseline. The investigators will study patients at baseline and at intervals On-Tx with teriflunomide in order to identify patients with active vs. stable disease, based on clinical (relapse) and radiological (new T2 hyperintense lesions) evidence. The investigators will study the expression of biomarkers in each patient subgroup.

C2. Primary endpoints. The central question of the study is whether the expression levels of one or more putative biomarker (TOB1, TLR2, TLR4, CCR1) differ(s) between patients from the two informative subgroups.

C3. Outcome measures. The outcomes that will address the central question of the study consist of the following:

1. Measures of protein expression levels of TLR2, TLR4 and CCR1 on CD4 T-subsets by flow cytometry.
2. TOB1 mRNA expression in CD4 T-subsets by quantitative RT-PCR (qRT-PCR) and the PrimeFlow RNA Assay.
3. Differences in mRNA or protein expression of selected markers in short-term cultures between patients from the two informative subgroups.

C4. Subject population. The study population includes:

1. treatment-naive patients with RRMS from the Montreal Neurological Hospital (MNH) MS clinics before treatment (pre-Tx) with teriflunomide; and
2. patients with RRMS that were previously treated with other disease modifiying therapies (DMTs) but that are switching to teriflunomide.

C5. Ethics approval: The study was approved by the Neurosciences Research Ethics Board of the MNH/MN. The data will be kept for 7 years.

C6. Consents. The Principal Investigator or his delegate will obtain informed consent

D. STUDY PROCEDURES. The study will investigate a biomarker signature in patients with MS who are being treated with teriflunomide by their neurologist.

D1. Participants and clinic visits. Before beginning treatment with teriflunomide, each patient will have a clinical evaluation, an MRI, as part of routine clinical practice, and a blood draw (see below). At intervals, participants will have a clinical evaluation and a second MRI evaluation to determine whether they have active vs. stable disease. In order to permit a phased approach, the neurologists will endeavor to identify patients after six months of treatment who show evidence of active vs. stable disease, approximately 3 in each subgroup. Blood draws will be obtained from each of these patients for subsequent laboratory studies (see below).

D2. Sample collection. Up to 120 ml of peripheral venous blood will be drawn from each subject at baseline and at intervals, to collect serum and plasma, to obtain total lymphocyte counts, CD3, CD4 and CD8 counts and to isolate peripheral blood mononuclear cells (PBMC) for immediate analysis and also for cryopreservation.

D3. Laboratory analysis.

D3.1. Naïve CD4 T-cell isolation and quantitative RT-PCR analysis of TOB1 expression. Reduced expression of TOB1, an inhibitor of T-cell proliferation, correlated with rapid progression from CIS to RRMS in one study (2), and also correlated in the investigators' previous study with rapid progression from RRMS to SPMS (2). The investigators will isolate naïve CD4 T-cells using MACS beads (2) and determine TOB1 expression by quantitative RT-PCR in a small cohort of patients (5-10 patients) and age-matched healthy controls (HCs).

D3.2. Analysis of cryopreserved PBMC.

Strategy 1. Surface protein expression of TLR2, TLR4 and CCR1 in CD4 T-subsets. The investigators will analyze baseline and On-Tx cryopreserved samples for expression (% positivity and MFI) of TLR2, TLR4 and CCR1 on naïve, central memory, effector memory, terminally differentiated effector memory and regulatory T-cells by flow cytometry on a BD LSRFortessa with a 5-laser system. The investigators will use FlowJo software for analysis. The investigators will identify the biomarker which is most informative, i.e. shows the greatest difference in expression levels between patients in the two informative subgroups at baseline or on treatment.

Strategy 2. Comparison of TOB1 mRNA expression by qRT-PCR and the PrimeFlow RNA Assay. The investigators will develop the PrimeFlow™ RNA assay (affymetrix Ebioscience) for simultaneous analysis of mRNA and protein expression. Initially, the investigators will compare TOB1 mRNA expression with that obtained by qRT-PCR, as qRT-PCR is the gold standard for mRNA quantification. The investigators will compare TOB1 mRNA expression in naïve CD4 T-cells by the two methods. If the measurements are comparable, the investigators will then be able to simultaneously assess TOB1 expression in naïve CD4 T-cells and the expression of the most informative biomarker in CD4 T-subsets and compare expression levels in patients from the two informative subgroups as outlined below.

Strategy 3. mRNA and protein kinetics of TOB1 and a T-cell biomarker in stimulated T-cells. The investigators anticipate that T-cell stimulation will identify differences between patients from the two informative subgroups in either mRNA or protein kinetics of TOB1 or one of our surface protein biomarkers. In other words, these studies may show differences between patients with active vs. stable MS.

This strategy involves a stimulation phase and an analytical phase as follows.

1. Firstly, after selecting patients from the two patient subgroups (3-4 patients/subgroup) and from age-matched HCs, the investigators will stimulate cryopreserved PBMC from baseline and one-year treatment samples using PMA/ionomycin and BD GolgiStop™ Protein Transport inhibitor for 4 hr at 37° C in 5% CO2. The investigators will determine the optimal concentrations of each reagent through assay-specific titration for use with the PrimeFlow RNA Assay.
2. The second phase will use the PrimeFlow RNA Assay to assess mRNA and protein kinetics of TOB1 and the most informative surface protein biomarker in patient subgroups and HCs. This assay can reveal the dynamics of both RNA and protein expression in individual cells and in T-subsets in response to T-cell stimulation. The utility of the PrimeFlow RNA assay was validated in a landmark study of T-subsets (4); detailed methods are available on the following website: http://www.ebioscience.com/media/newpdf/PrimeFlowRNAAssayUM010915.pdf.

D4. Statistical analysis. The investigators will use GraphPad Prism 7 for all statistical analyses, and use appropriate parametric or non-parametric tests according to the data distribution.

E. ANTICIPATED RESULTS. Firstly, the investigators anticipate that one or more T-subsets in baseline PBMC samples (before teriflunomide treatment) will show increased surface protein expression of one or more T-cell activation molecules in the patients that show disease activity On-Tx vs. patients that do not show disease activity On-Tx. Such a finding may help identify patients for whom teriflunomide is the optimal DMT. Secondly, treatment with teriflunomide may alter the expression of one or more T-cell activation molecules in one or more T-subsets and this alteration may correlate with reduced disease activity, thereby suggesting that altered T-cell activation contributes to a positive response to teriflunomide. Thirdly, short term cultures of baseline samples vs. one-year samples from patients and from age-matched HCs may identify differences in mRNA and protein kinetics of a T-cell activation marker in patients at baseline, which then revert to a normal pattern in those with no disease activity at one year. Such findings would point towards important functional alterations mediated by teriflunomide that correlate with a positive therapeutic response.

F. STUDY SITES All patients will be recruited from the Montreal Neurological Hospital MS Clinics and all experimental work will be done in the Duff Medical Building, Department of Pathology, McGill University.

G. TIMELINES G.1. First Patient In (FPI) - one month after execution of the contract and ethics approval.

G.2. Last Patient In (LPI) ~ 12-15 months after execution of the contract and ethics approval: this reflects the time required to recruit a total of up to 75 patients treated withTeriflunomide.

G.3. Interim analyses

* Assess recruitment rate at 2 months to consider inclusion of satellite centers.
* RT-PCR analysis of TOB1 in 5-10 patients Pre-TX and age-matched HCs (4 months).
* Preliminary flow cytometry analysis of surface protein biomarkers based on the tentative identification of ~ 3 active vs. ~ 3 stable patients identified at the 8 month On-Tx time point
* Additional flow cytometry analysis of surface protein biomarkers on a further 3 active vs. 3 stable patients identified at the 14 month On-Tx time point.

G4. Progress Reports. Quarterly progress updates on patient recruitment and biannual report on clinical evaluation parameters to subgroup patients.

G5. Last Patient Visit (LPLV) - 24-27 months. G6. Completion of Final Report - 30 months. G7. Projected Manuscript Submission. 33 months. H. APPENDICES APPENDIX 1. Primary Antibody Panel

1. FVS 510 (BD)
2. CD4 BUV395 (BD)
3. CD45RA BV421 (BD)
4. CD127 BUV737 (BD)
5. CD25 BV786 (BD)
6. CCR1 Alexa Fluor® 488 (R&D Sys.)
7. TLR2 PE (eBioscience)
8. CCR7 PE-CF594 (BD)
9. CD14 PerCP-Cy5.5 (BD)
10. TLR4 APC (eBioscience)
11. CD3 APC-H7 (BD) FVS 510: BD Horizon™ Fixable Viability Stain 510 BUV: BD Horizon™ Brilliant Ultraviolet™ BV: BD Horizon™ Brilliant Violet™ Alexa Fluor® (Molecular Probes) (sometimes abbrev. AF) PE-CF594: BD Horizon™ PE-CF594 APC-H7: BD Pharmingen™ APPENDIX 2. PrimeFlow™ RNA Assay Panels including TLR2 as a possible biomarker - under development

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive patients with relapsing-remitting multiple sclerosis
* Patients treated previously with one or more previous disease-modifying treatments but with a washout period of at least 4 weeks before starting treatment with teriflunomide.

Exclusion Criteria:

* Acute infections in the preceding 4 weeks
* Vaccination in the previous 2 months
* An active malignancy (except basal cell carcinoma)
* Pregnant or breastfeeding patients
* Communication difficulty, i.e. unable to understand the study
* Vulnerable patients, i.e. unable to provide informed consent or lacking legal freedom, e.g. prisoners

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with relapsing-remitting MS who agree to be treated with teriflunomide
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Biomarkers and disease activity in patients treated with Teriflunomide (Aubagio) | 26 months
  Primary outcome measure
  * Membrane expression of TLR2, TLR4 and CCR1 Percent expression and mean fluorescence intensity in CD4 T-cell subsets in active vs. stable patient groups
  * TOB1 expression by real-time PCR on CD4 T-cell subsets Number of molecules per µg cDNA
  * PrimeFLow assay Number of T-cells expressing both mRNA and surface membrane TLR2 Number of T-cells expressing mRNA for TOB1 Number of T-cells expressing mRNA for TOB 1 and surface protein for TLR2

CONTACTS AND LOCATIONS:
Overall Officials: David Haegert, MD, Principal Investigator — McGill University
Locations (1):
- Department of Pathology, Montreal, Quebec, Canada

REFERENCES:
- [Background] Kieseier BC, Wiendl H. New evidence for teriflunomide in multiple sclerosis. Lancet Neurol. 2014 Mar;13(3):234-5. doi: 10.1016/S1474-4422(14)70012-2. Epub 2014 Jan 23. No abstract available. PMID 24461573
- [Background] Zastepa E, Fitz-Gerald L, Hallett M, Antel J, Bar-Or A, Baranzini S, Lapierre Y, Haegert DG. Naive CD4 T-cell activation identifies MS patients having rapid transition to progressive MS. Neurology. 2014 Feb 25;82(8):681-90. doi: 10.1212/WNL.0000000000000146. Epub 2014 Jan 22. PMID 24453076
- [Background] Corvol JC, Pelletier D, Henry RG, Caillier SJ, Wang J, Pappas D, Casazza S, Okuda DT, Hauser SL, Oksenberg JR, Baranzini SE. Abrogation of T cell quiescence characterizes patients at high risk for multiple sclerosis after the initial neurological event. Proc Natl Acad Sci U S A. 2008 Aug 19;105(33):11839-44. doi: 10.1073/pnas.0805065105. Epub 2008 Aug 8. PMID 18689680
- [Background] Porichis F, Hart MG, Griesbeck M, Everett HL, Hassan M, Baxter AE, Lindqvist M, Miller SM, Soghoian DZ, Kavanagh DG, Reynolds S, Norris B, Mordecai SK, Nguyen Q, Lai C, Kaufmann DE. High-throughput detection of miRNAs and gene-specific mRNA at the single-cell level by flow cytometry. Nat Commun. 2014 Dec 4;5:5641. doi: 10.1038/ncomms6641. PMID 25472703